CLINICAL TRIAL: NCT03550209
Title: Fatty Acid Supplements Alter Biological Signatures in Children With Autism Spectrum Disorder
Brief Title: Fatty Acid Supplementation in Children With ASD
Acronym: Omega Heroes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarah Keim (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Sarah Keim, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB17-00517; R61AT009632 (NIH)
Record Dates: First submitted 2018-05-24; First posted 2018-06-08 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LCPUFA Oil Supplement, Low Dose (Experimental): 25 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  Interventions: Drug: LCPUFA Oil Supplement
- LCPUFA Oil Supplement, Medium Dose (Experimental): 50 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  Interventions: Drug: LCPUFA Oil Supplement
- LCPUFA Oil Supplement, High Dose (Experimental): 75 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  Interventions: Drug: LCPUFA Oil Supplement
- Canola Oil (Placebo Comparator): Equal volume (25 mg/kg, 50 mg/kg, or 75 mg/kg) of placebo (canola) oil to be administered twice per day by mouth for 90 days
  Interventions: Dietary Supplement: Canola Oil Placebo

INTERVENTIONS:
Drug: LCPUFA Oil Supplement — 25 mg/kg, 50 mg/kg, or 75 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  Arms: LCPUFA Oil Supplement, High Dose; LCPUFA Oil Supplement, Low Dose; LCPUFA Oil Supplement, Medium Dose
Dietary Supplement: Canola Oil Placebo — Equal volume (25 mg/kg, 50 mg/kg, or 75 mg/kg) of placebo (canola) oil to be administered twice per day by mouth for 90 days
  Arms: Canola Oil

SUMMARY:
The purpose of this study is to examine how fatty acid supplementation alters biological signatures in children with ASD

DETAILED DESCRIPTION:
Children with Autism Spectrum Disorder (ASD) suffer from both mental and physical symptoms that affect their quality of life and severely disrupt family well-being. Fatty acid supplements are natural products with anti-inflammatory properties often used for treatment of ASD symptoms, but their efficacy remains unproven. The objective of the proposed protocol is to quantify the impact of Omega 3-6 on pre-specified biological signatures. The hypotheses were formulated based on data from the investigators previous studies and other published data which suggest that the inflammatory markers, IL-1β, IL-2, and IFNγ are consistently elevated in children with ASD and decreases in these markers correlate with ASD symptom improvement. The investigators long-term goal is to identify effective treatments for ASD.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-6 years old
* ASD diagnosis at Nationwide Children's Hospital within the prior 6 months
* ADOS-2 score in "autism" (severe) range
* English is primary language

Exclusion Criteria:

* Fatty acid supplementation in the past 6 months
* Consumes fatty fish more than 3 times per week
* Still breastfeeding or formula feeding
* Quadriparesis
* Deafness
* Blindness
* Seizure disorder diagnosis
* Autoimmune disorder including Type 1 Diabetes, Fragile X, Rett, Angleman Syndromes, Tuberous Schlerosis
* Feeding problems precluding consumption of the supplement
* Ingredient allergy (canola, fish, or borage seed)
* Planned surgeries scheduled within the time frame of trial participation

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Keim, PhD, Principal Investigator — Nationwide Children's Hospital; Lynette Rogers, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Keim SA, Jude A, Smith K, Khan AQ, Coury DL, Rausch J, Udaipuria S, Norris M, Bartram LR, Narayanan AR, Rogers LK. Randomized Controlled Trial of Omega-3 and -6 Fatty Acid Supplementation to Reduce Inflammatory Markers in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2022 Dec;52(12):5342-5355. doi: 10.1007/s10803-021-05396-9. Epub 2022 Jan 11. PMID 35013866

RESULTS

PARTICIPANT FLOW:
Groups:
- LCPUFA Oil Supplement, Low Dose: 25 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  LCPUFA Oil Supplement: 25 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
- LCPUFA Oil Supplement, Medium Dose: 50 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  LCPUFA Oil Supplement: 50 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
- LCPUFA Oil Supplement, High Dose: 75 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
  LCPUFA Oil Supplement: 75 mg/kg of GLA+EPA+DHA as Omega 3-6 oil to be administered twice per day by mouth for 90 days
- Canola Oil: Equal volume of placebo (canola) oil to be administered twice per day by mouth for 90 days
  Canola Oil Placebo: Equal volume of placebo (canola) oil to be administered twice per day by mouth for 90 days
Period: Overall Study
Arm/Group | LCPUFA Oil Supplement, Low Dose | LCPUFA Oil Supplement, Medium Dose | LCPUFA Oil Supplement, High Dose | Canola Oil
Started | 12 | 12 | 13 | 35
Completed | 11 | 9 | 11 | 31
Not Completed | 1 | 3 | 2 | 4
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 2
Not completed — Excluded due to ineligibility after randomization | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 72 participants were randomized into the study, but only 70 participants were included in analysis. Two participants who were randomized to receive canola oil (placebo) were found to be ineligible after randomization. These two participants were unenrolled from the study by the Principal Investigators and were not included in any analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCPUFA Oil Supplement, Low Dose | LCPUFA Oil Supplement, Medium Dose | LCPUFA Oil Supplement, High Dose | Canola Oil | Total
Number analyzed (Participants) | 12 | 12 | 13 | 33 | 70
Age, Customized [Count of Participants; unit: Participants]
  2-3 years | 7 | 7 | 7 | 15 | 36
  4-6 years | 5 | 5 | 6 | 18 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 5 | 13
  Male | 9 | 10 | 10 | 28 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 2 | 6
  Not Hispanic or Latino | 11 | 9 | 13 | 31 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African-American | 4 | 2 | 4 | 3 | 13
  Race: White | 6 | 6 | 8 | 27 | 47
  Race: Other or Multiple Races | 2 | 3 | 1 | 3 | 9
  Race: Missing | 0 | 1 | 0 | 0 | 1
Baseline Pre-Specified Biological Signatures (cytokines) [Mean (Standard Deviation); unit: pg/ml] — A blood draw was completed at the first study visit prior to beginning any study interventions. This blood draw was used to collect baseline data for pre-specified biological signatures.
  pg/ml
    IL-1β | 0.10 (0.05) | 0.16 (0.25) | 0.07 (0.05) | 0.10 (0.06) | 0.11 (0.04)
    IL-2 | 0.31 (0.12) | 0.55 (0.96) | 0.23 (0.10) | 0.48 (0.47) | 0.39 (0.15)
    IFNγ | 8.95 (6.40) | 11.22 (10.18) | 9.80 (7.35) | 16.72 (43.17) | 11.67 (3.49)

OUTCOME MEASURES:

1. Primary Outcome: Bioavailability
Description: Group differences in bioavailability; each fatty acid as a percent of total erythrocyte fatty acids at the end of the trial
Time Frame: Baseline to 90 days post-randomization
Population: 11 participants were not included in analysis due to missing a scheduled blood draw at 90 days post randomization.
Measure: Mean (Standard Deviation); unit: mol%
Arm/Group | LCPUFA Oil Supplement, Low Dose | LCPUFA Oil Supplement, Medium Dose | LCPUFA Oil Supplement, High Dose | Canola Oil
Number analyzed (Participants) | 9 | 9 | 11 | 30
mol%
  EPA | 1.95 (1.04) | 1.80 (1.56) | 3.00 (2.45) | 0.80 (0.33)
  DHA | 4.33 (1.26) | 3.61 (1.39) | 4.75 (1.76) | 2.46 (0.92)

2. Primary Outcome: Safety (Adverse Events)
Description: Average number of adverse events per treatment group
Time Frame: Baseline to 90 days post-randomization
Measure: Mean (Standard Deviation); unit: events per person
Arm/Group | LCPUFA Oil Supplement, Low Dose | LCPUFA Oil Supplement, Medium Dose | LCPUFA Oil Supplement, High Dose | Canola Oil
Number analyzed (Participants) | 12 | 12 | 13 | 33
events per person | 4.5 (2.35) | 3.33 (2.23) | 5.62 (2.81) | 3.88 (2.53)

3. Primary Outcome: Biological Signatures
Description: Changes in the biological signatures (IL-1β, IL-2, IFNγ) from baseline to the end of the trial.
Time Frame: Baseline to 90 days post-randomization
Population: 11 participants were not included in analysis due to missing a scheduled blood draw at 90 days post randomization.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | LCPUFA Oil Supplement, Low Dose | LCPUFA Oil Supplement, Medium Dose | LCPUFA Oil Supplement, High Dose | Canola Oil
Number analyzed (Participants) | 9 | 9 | 11 | 30
pg/ml
  IL-1β | -0.01 (0.64) | -0.02 (0.38) | -0.03 (0.16) | 0.11 (0.09)
  IL-2 | -0.10 (0.34) | -0.29 (0.01) | -0.11 (0.26) | 0.01 (0.24)
  IFNγ | -1.04 (0.67) | -1.43 (0.56) | 2.99 (0.19) | -9.77 (43.92)

ADVERSE EVENTS:
Time Frame: Baseline to 90 days post-randomization
Arm/Group | LCPUFA Oil Supplement, Low Dose | LCPUFA Oil Supplement, Medium Dose | LCPUFA Oil Supplement, High Dose | Canola Oil
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/33
Other Adverse Events (participants affected / at risk) | 12/12 | 11/12 | 13/13 | 31/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCPUFA Oil Supplement, Low Dose (N=12) | LCPUFA Oil Supplement, Medium Dose (N=12) | LCPUFA Oil Supplement, High Dose (N=13) | Canola Oil (N=33)
Ear (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 3 (4) | 6 (6) — Includes ear infection, poor hearing, and fluid in ears.
Eye (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) — Includes eye irritation and conjunctivitis.
Gastrointestinal (Gastrointestinal disorders) | 8 (16) | 10 (14) | 12 (30) | 22 (38) — Includes changes in appetite, constipation, diarrhea, stomach pain/discomfort, changes in frequency of bowel movements, flatulence, heartburn, changes in stool color/consistency, vomiting, and gastrointestinal virus.
Infectious (Infections and infestations) | 5 (7) | 4 (4) | 8 (9) | 19 (21) — Includes common cold, fever, feeling flushed/warm, flu, and hand, foot and mouth.
Accidental Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 2 (2) — Includes head injury, chin laceration, etc.
Muscular (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (4) — Includes muscle, joint and bone pain, head shaking, clumsiness, improved motor skills, and tics.
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Psychological (Psychiatric disorders) | 5 (6) | 4 (5) | 7 (9) | 12 (17) — Includes anxiety, aggression, increase in negative behaviors/emotions, confusion/slowed thinking, irritability, changes with speech, better memory, and understanding more.
Genital (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Includes diurnal enuresis and improved toilet training.
Nose (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3) | 4 (5) | 4 (5) — Includes nasal/sinus congestion, runny nose, sore throat, strep throat, and tonsillectomy.
Skin (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 2 (2) | 6 (7)
Mouth (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) — Includes teething and jaw pain.
Chest (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6) | 5 (5) | 9 (9) — Includes allergies, bronchitis, cold symptoms, coughing, and upper respiratory infection.
Energy (Nervous system disorders) | 3 (3) | 2 (3) | 0 (0) | 4 (4) — Includes overly excited or energetic, calmness, and fatigue.
Sleep (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 6 (6) — Includes difficulty falling asleep, interrupted sleep, nightmares, drowsiness, and sleeping too much.

LIMITATIONS AND CAVEATS:
There were initially unanticipated obstacles in identifying enough patients because the ADOS scores were not consistently available for all patients in the electronic medical record system (EPIC), and this score served as part of the eligibility criteria. This problem was solved, and our recruitment pace rebounded, we went from approximately 2-3 enrollments per month to 6.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03550209/Prot_SAP_002.pdf
  • Informed Consent Form (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT03550209/ICF_001.pdf